CLINICAL TRIAL: NCT01893593
Title: A Cluster Randomized Trial of the Implementation of the NHLBI Expert Panel Integrated Guidelines for Cardiovascular Health and Risk Reduction in Children and Adolescents
Brief Title: Young Hearts, Strong Starts
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: RTI International (Other)
Collaborators: East Carolina University (Other); Pediatric Practice Research Group (Network); Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Young Hearts, Strong Starts
Record Dates: First submitted 2013-06-27; First posted 2013-07-09 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Cardiovascular Risk Reduction
Keywords: Cardiovascular risk; lifestyle change; blood pressure; body mass index; tobacco
MeSH Terms: interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Other): Usual care
  Interventions: Other: Control
- Intervention (Active Comparator): Multifaceted intervention to improve clinical systems
  Interventions: Other: Intervention

INTERVENTIONS:
Other: Intervention — Guideline summary and data feedback from a baseline medical record review and a multifaceted intervention to improve clinical systems
  Arms: Intervention
Other: Control — Guideline summary and data feedback from a baseline medical record review
  Arms: Control

SUMMARY:
This is a cluster randomized trial of pediatric cardiovascular risk reduction guideline implementation in 32 clinical practices

DETAILED DESCRIPTION:
Objective: The Young Hearts Strong Starts Study was designed to test strategies to facilitate adoption of the Integrated Guidelines for Cardiovascular Health and Risk Reduction in Children and Adolescents among pediatric and family medicine providers. The study compares quality measures based on the guidelines for two dissemination strategies: a multi-faceted, practice-directed intervention or standard dissemination.

Methods: Two primary care research networks recruited practices and provided support for the intervention and outcome evaluations. Individual practices were randomly assigned to either the intervention or control groups using a cluster randomized design based on network affiliation, number of clinicians per practice, urban vs. nonurban location, and practice type. In this design, the units of observation are individual children because outcomes are abstracted from medical records for individual patients. The units of randomization are physician practices. This results in a multilevel design in which patients are nested within practices. Implementation The intervention practices receive toolkits, including guideline summaries and slides, a patient and family behavior change workbook, and a clinical decision support tool. Guideline implementation was promoted through an introductory academic detailing session and the use of an ongoing e-learning group. The intervention strategy was further enhanced by aligning this project with the American Board of Pediatrics quality improvement Maintenance of Certification (MOC) requirements and offers voluntary MOC participation to participants. MOC participation includes the creation of a practice aims statement, monthly physician self-abstraction to track progress throughout the intervention, and participation in webinar presentations and sharing of best practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients seen for well child visits

Exclusion Criteria:

* Terminally ill patients

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2011-11; Primary Completion 2012-12 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Summary composite measure of practice performance and exposure | One year
  Summary measures of the number of guideline recommended actions in each area divided by the number of eligible patients. Process measures of adherence to guidelines in the measurement, interpretation, and recommendations for blood pressue and BMI, and measures of assessment and advice for tobacco exposure and use.

SECONDARY OUTCOMES:
Measures of guideline adherence for BMI, blood pressure, and tobacco use and exposure | One year
  Process measures of adherence to guidelines in the measurement, interpretation, and recommendations for blood pressue and BMI, and measures of assessment and advice for tobacco exposure and use.

CONTACTS AND LOCATIONS:
Overall Officials: Ken LaBresh, MD, Principal Investigator — RTI International
Locations (2):
- United States (2):
  - Lurie Children's Hospital, Chicago, Illinois
  - East Carolina University, Greenville, North Carolina

REFERENCES:
- [Derived] LaBresh KA, Ariza AJ, Lazorick S, Furberg RD, Whetstone L, Hobbs C, de Jesus J, Salinas IG, Bender RH, Binns HJ. Adoption of cardiovascular risk reduction guidelines: a cluster-randomized trial. Pediatrics. 2014 Sep;134(3):e732-8. doi: 10.1542/peds.2014-0876. PMID 25157013
- [Derived] LaBresh KA, Lazorick S, Ariza AJ, Furberg RD, Whetstone L, Hobbs C, de Jesus J, Bender RH, Salinas IG, Binns HJ. Implementation of the NHLBI integrated guidelines for cardiovascular health and risk reduction in children and adolescents: rationale and study design for young hearts, strong starts, a cluster-randomized trial targeting body mass index, blood pressure, and tobacco. Contemp Clin Trials. 2014 Jan;37(1):98-105. doi: 10.1016/j.cct.2013.11.011. Epub 2013 Dec 1. PMID 24295879